CLINICAL TRIAL: NCT07239271
Title: A Multicenter Phase III Clinical Study and Translational Research on Adaptive Neoadjuvant Therapy of De-escalation and Escalation for HER2-Positive Breast Cancer Based on Multi-Omics Response Evaluation Model
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ma Fei，MD, Chief Physician, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC5389
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-06

CONDITIONS: Patients With HER2-positive Breast Cancer (BC) Suitable for Neoadjuvant Therapy

STUDY DESIGN:
Intervention Model Description: This is a multicenter, prospective, randomized phase III clinical trial, planning to enroll 2,000 subjects (1:3 randomized control grouping, 500 in the control group, 1,500 in the experimental group).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- The control group received the TCbHP regimen (Active Comparator): The control group received the TCbHP regimen (docetaxel, carboplatin, trastuzumab, and pertuzumab)
  Interventions: Drug: The control group
- Adaptive therapy of de-escalation and escalation based on imaging and molecular Analysis (Experimental): At baseline, patients receive the Nab-P+HP regimen (albumin-bound paclitaxel plus trastuzumab and pertuzumab).After one cycle of treatment (C1), ctDNA testing is performed. After two cycles of treatment , radiological evaluation is conducted. If the patient is ctDNA (-) and achieves PR, they continue with the Nab-P+HP regimen . If the patient is ctDNA (-) and non-PR, they receive the TCbHP regimen for two cycles. If the patient is ctDNA (+) and has no mutations in the PI3K/AKT/mTOR (PAM)pathway, they receive the PyroHT regimen (pyrotinib plus trastuzumab and docetaxel) for two cycles. If the patient is ctDNA (+) at baseline or after one treatment cycle and has PAM pathway mutations, they receive the EveroHT regimen (everolimus plus trastuzumab and docetaxel) for two cycles. If the patient achieves PR after C4, they continue with the regimen for another two cycles. If PR is not achieved，the patient switches to ADC or AC+H (anthracycline plus cyclophosphamide plus trastuzumab) regimen
  Interventions: Drug: Adaptive therapy of de-escalation and escalation based on imaging and molecular analysis for predicting response

INTERVENTIONS:
Drug: The control group — received the TCbHP regimen (docetaxel, carboplatin, trastuzumab, and pertuzumab)
  Arms: The control group received the TCbHP regimen
Drug: Adaptive therapy of de-escalation and escalation based on imaging and molecular analysis for predicting response — At baseline, patients receive the Nab-P+HP regimen (albumin-bound paclitaxel plus trastuzumab and pertuzumab).After one cycle of treatment (C1), ctDNA testing is performed. After two cycles of treatment , radiological evaluation is conducted. If the patient is ctDNA (-) and achieves PR, they continue with the Nab-P+HP regimen . If the patient is ctDNA (-) and non-PR, they receive the TCbHP regimen for two cycles. If the patient is ctDNA (+) and has no mutations in the PI3K/AKT/mTOR (PAM)pathway, they receive the PyroHT regimen (pyrotinib plus trastuzumab and docetaxel) for two cycles. If the patient is ctDNA (+) at baseline or after one treatment cycle and has PAM pathway mutations, they receive the EveroHT regimen (everolimus plus trastuzumab and docetaxel) for two cycles. If the patient achieves PR after C4, they continue with the regimen for another two cycles. If PR is not achieved，the patient switches to ADC or AC+H (anthracycline plus cyclophosphamide plus trastuzumab) regimen
  Arms: Adaptive therapy of de-escalation and escalation based on imaging and molecular Analysis

SUMMARY:
This study is a phase III clinical trial to explore the efficacy and safety of HER2-positive breast cancer neoadjuvant adaptive therapy compared with standard therapy based on multi-omics data, and to explore a new prediction model for pCR. The trial protocol in this study design has sufficient preliminary basis.

HER2-targeted therapies can significantly improve pCR rates and enhance clinical outcomes in HER2-positive breast cancer patients undergoing neoadjuvant treatment. However, standard neoadjuvant regimens typically involve multiple chemotherapeutic agents, often accompanied by severe adverse reactions. To optimize neoadjuvant strategies, minimize chemotherapy-related toxicities, and maximize the therapeutic advantages of anti-HER2 therapies, research on downstaging chemotherapy regimens has been intensively pursued. The first phase III HELEN-006 study evaluating the efficacy and safety of albumin-bound paclitaxel combined with neoadjuvant chemotherapy (nab-PHP) in HER2-positive breast cancer, led by Professor Liu Zhenzhen's team at Henan Cancer Hospital, was published online in The Lancet Oncology. This landmark study demonstrated that the nab-PHP regimen achieved higher pCR rates and better tolerability compared to the standard TCbHP regimen, charting a new course for downstaging chemotherapy approaches.

In recent years, new anti-HER2 drugs such as pyrotinib, T-DM1, and T-DXd have been continuously developed and launched, achieving good results in the treatment of HER2-positive breast cancer. These advances have changed clinical practice and are recommended in domestic and international guidelines for second-line or later-line treatment of advanced HER2-positive breast cancer. Their efficacy in neoadjuvant therapy is still being explored. The PHEDRA study is a multicenter, double-blind, randomized, controlled phase 3 trial that included a total of 355 patients: 178 in the group receiving docetaxel and trastuzumab combined with pyrotinib (TH+Py), and 177 in the group receiving docetaxel and trastuzumab combined with placebo. The study results show that the pCR rate in the TH+Py group was significantly higher than in the TH+placebo group (41.0% vs. 22.0%, P<0.0001). The DESTINY-Breast 11 study is an open-label phase III clinical trial designed to investigate the efficacy and safety of neoadjuvant T-DXd monotherapy or T-DXd followed by sequential THP compared with dose-dense doxorubicin and cyclophosphamide followed by sequential THP (ddAC-THP) in patients with high-risk, early-stage HER2+ breast cancer. Patients with locally advanced HER2+ breast cancer, either HR+ or HR-, were randomized in a 1:1:1 ratio to Group A (T-DXd monotherapy), Group B (T-DXd followed by sequential THP), or Group C (ddAC-THP). The primary endpoint is pathological complete response (pCR). Currently, the DESTINY-Breast 011 study is still ongoing. At the 2024 SABCS conference, results were reported from a prospective, randomized, open-label phase II trial of SHR-A1811, a HER2-targeted antibody-drug conjugate, in the neoadjuvant treatment of HER2-positive early breast cancer. The main goal of this study is to assess the efficacy and safety of SHR-A1811 in the neoadjuvant treatment of HER2-positive early breast cancer. Open-label, phase II trial; the primary objective of this study is to explore the efficacy and safety of SHR-A1811 as neoadjuvant therapy in HER2-positive early-stage breast cancer. The pCR rate of SHR-A1811 monotherapy was 63.2% in the overall population, 50.0% in HR+ breast cancer, and 74.5% in HR- breast cancer. Everolimus is an mTOR inhibitor that can suppress the "phosphatidylinositol 3-kinase/protein kinase B/mammalian target of rapamycin (PI3K/Akt/mTOR)" signaling pathway in tumor cells, thereby exerting an anti-cancer effect. In the BOLERO-3 clinical study, for patients with advanced disease who had failed anti-HER2 therapy, adding everolimus to vinorelbine plus trastuzumab prolonged the duration of disease control by about 1.2 months.

Our research group has previously established a nationwide multicenter multi-omics database that includes clinical information, pathological characteristics, and ctDNA data from 958 patients with advanced breast cancer. This has clarified the gene mutation profiles and prognostic features of advanced breast cancers with different molecular subtypes. Subsequently, we further developed a dynamic ctDNA monitoring sample library with 430 cases, tracking gene changes at multiple time points during the treatment of advanced breast cancer patients. By integrating clinical information, pathological features, and other multi-omics data, we comprehensively explored the process of tumor clonal evolution during treatment in patients with advanced breast cancer, providing a solid foundation for the development of efficacy prediction models.

This study is a nationwide, multicenter, prospective, randomized, controlled phase III clinical trial. It aims to compare the efficacy and safety of mu

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 18-70 years;
2. ECOG Performance Status (PS) score of 0-1;
3. Histologically confirmed operable early or locally advanced invasive breast cancer, with a primary tumor diameter >2 cm;
4. Patients with pathologically or cytologically confirmed primary breast cancer. For multifocal tumors (multiple tumors confined to the same quadrant as the primary tumor), it is recommended that all lesions be confirmed as HER2-positive prior to enrollment;
5. TNM stage II-IIIc (T2-3, N0-1, M0 or T2-3, N2-3, M0 or T4, any N, M0);
6. Pathologically confirmed HER2 positivity: IHC result of 3+ or 2+/ISH+;
7. Known status of estrogen receptor (ER), progesterone receptor (PgR), and Ki-67;
8. The patient agrees to provide tumor tissue and blood samples as specified in the protocol;
9. It is recommended that the patient's organ function meets the following requirements, as determined by the investigator based on each patient's condition:

   1. Complete blood count (no blood transfusion within the past 14 days): Neutrophils (ANC) ≥1.5×10⁹/L; Platelets (PLT) ≥100×10⁹/L; Hemoglobin (Hb) ≥90 g/L; White blood cells (WBC) ≥2.5×10⁹/L;
   2. Blood biochemistry: Total bilirubin (TBIL) ≤1.5 times the upper limit of normal (ULN); for patients with Gilbert's syndrome, TBIL ≤2×ULN; Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN; Creatinine (Cr) ≤1.5×ULN;
   3. Coagulation tests must meet the following criteria: Prothrombin time (PT), activated partial thromboplastin time (APTT), and international normalized ratio (INR) ≤1.5×ULN (for patients not on anticoagulation); for patients on anticoagulation, PT within the expected range for prescribed anticoagulants is acceptable;
   4. Cardiac echocardiography: Left ventricular ejection fraction (LVEF) ≥55%;
10. Preoperative assessment indicates that the patient is likely to meet the surgical criteria after neoadjuvant therapy, is able to undergo surgery as assessed by the investigator, and can receive adjuvant therapy after surgery;
11. Non-lactating women with a negative serum or urine pregnancy test within 7 days prior to enrollment; women of childbearing potential must agree to use highly effective contraception during the study and for 6 months after the last dose of study medication;
12. Expected survival of more than 3 months;
13. The subject voluntarily agrees to participate in this study, signs an informed consent form, and demonstrates good compliance.

Exclusion Criteria:

1. Patients with metastatic breast cancer;
2. Patients with multifocal tumors (tumors involving more than one quadrant) or bilateral breast cancer;
3. Patients with a history of prior anti-tumor treatment, such as chemotherapy, endocrine therapy, HER2-targeted biological therapy, or previous breast surgery (excluding diagnostic biopsy for primary breast cancer);
4. Patients who have had or currently have other malignant tumors within the past 3 years. The following two situations are exceptions and may be included: other malignancies treated by a single operation and have achieved 5 consecutive years of disease-free survival (DFS); cured carcinoma in situ of the cervix, non-melanoma skin cancers, and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ), and T1 (tumor invades lamina propria)];
5. Patients currently receiving treatment in other clinical studies (except those in overall survival follow-up in another study);
6. Patients who received major surgery, incisional biopsy, or significant traumatic injury within 28 days prior to initiation of study treatment (excluding diagnostic biopsy for primary breast cancer);
7. Patients with long-term non-healing wounds or fractures;
8. Patients with a history of substance abuse who are unable to abstain, or those with psychiatric disorders;
9. Subjects with any serious and/or uncontrolled diseases, including:

   1. History of hypertensive crisis or hypertensive encephalopathy, or uncontrolled hypertension (systolic blood pressure >150 mmHg or diastolic blood pressure >100 mmHg after antihypertensive treatment);
   2. History of heart failure or systolic dysfunction (LVEF < 55%);
   3. Myocardial ischemia or myocardial infarction of grade ≥2, arrhythmias (including male QTc≥450 ms, female QTc≥470 ms), and congestive heart failure of grade ≥2 (New York Heart Association [NYHA] classification);
   4. Angina pectoris requiring anti-anginal medication;
   5. Clinically significant heart valve disease;
   6. Positive screening for HCV, HIV, specific antitreponemal antibody, HBsAg, and peripheral blood HBV DNA level exceeding the normal range;
10. Imaging (CT or MRI) shows tumor invasion of major blood vessels, or in the investigator's judgment the tumor is highly likely to invade major vessels and cause fatal hemorrhage during the study;
11. History of active autoimmune disease requiring systemic treatment (e.g., with disease-modifying drugs, corticosteroids or immunosuppressants) within 2 years prior to study treatment initiation. Replacement therapy (e.g., thyroxine, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency) is not considered systemic treatment;
12. Diagnosed with immunodeficiency or receiving systemic glucocorticoid treatment or any other form of immunosuppressive therapy (dose >10 mg/day prednisone or equivalent), and continues to use it within 2 weeks prior to first dosing;
13. Other comorbidities that would interfere with the planned treatment, including severe pulmonary dysfunction/disease, active or uncontrolled severe infection (≥CTCAE 5.0 grade 2 infection);
14. Allergic to any component or excipient of the study drug(s);
15. Participation in other anti-tumor drug clinical trials within 4 weeks prior to randomization;
16. Pregnant or breastfeeding women, women of childbearing potential with a positive baseline pregnancy test, or women of childbearing age unwilling to use effective contraception throughout the study;
17. In the investigator's opinion, patients with concomitant diseases that seriously endanger subject safety or affect study completion, or for any other reason are deemed unsuitable for enrollment.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 2000 (Estimated)
Dates: Start 2025-11-16 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate | 2 year
  the proportion of patients assessed as having a pathological complete response after surgery among all patients who underwent surgery.

SECONDARY OUTCOMES:
Objective response rate | 2 year
  The proportion of patients whose tumors have shrunk to a certain standard and maintained that reduction for a period of time, including cases of CR and PR. Tumor objective response is evaluated using the Response Evaluation Criteria in Solid Tumors (RECIST 1.1).
3-year EFS rate | 3 year
  3-year event-free survival rate (3-year EFS rate): defined as the survival rate of all patients who have not experienced the expected endpoint event from randomization to the third year
3-year invasive disease-free survival rate | 3 year
Breast Conservation Rate | 2 years
Patient Report Outcomes | 2 years
  Assessed using the Breast Cancer Patient-Reported Outcome (PRO) scale 1.0 (NCC-BC-A 1.0)

IPD SHARING:
Plan to Share IPD: Undecided